CLINICAL TRIAL: NCT05954455
Title: Exploring Bulbar Function, Speech And Communication Development in SMA Type 1 (ExSpAnD SMA)
Brief Title: Exploring Bulbar Function, Speech And Communication Development in SMA Type 1
Acronym: ExSpAnD SMA
Status: Recruiting | Type: Observational
Sponsor: Institute of Child Health (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19NM18
Record Dates: First submitted 2023-06-29; First posted 2023-07-20 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: SMA1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
5q-spinal muscular atrophy (5q-SMA) is a rare, autosomal recessive neuromuscular disease characterized by degeneration of motor neurons in the spinal cord and lower brainstem with progressive muscle atrophy, weakness, and paralysis. The incidence is 1 in 7-10,000 live births. 5q-SMA presents a wide range of phenotypes that are classified into five clinical groups depending on age of onset and maximum motor milestone achieved. SMA type 1 presents shortly after birth and before six months of age with inability to achieve independent sitting and limited life expectancy due to respiratory complications (high mortality rate by 2 years of age). In addition to the severe gross-motor and respiratory impairment, bulbar weakness and dysfunction represent an obstacle to the development of verbal skills in these patients. To date, very little is known about these functions in children with SMA 1. With the increasing number of long-term SMA 1 survivors worldwide thanks to the availability of new pharmacological treatments, it has become obvious that treated children show new phenotypes, presenting changes not only in motor and respiratory function, but also in other domains, including bulbar function, speech and communication development. We aim to investigate the evolution of bulbar function and speech/communication development in children with SMA type 1 treated with approved disease-modifying therapies through validate scales and questionnaires for the paediatric population. Additional neurophysiological and neuroimaging studies will be offered on an optional basis to further investigate the underlying brain electrical activity, and brain structural and functional organization. The information gathered would promote the definition of additional outcome measures capturing improvement at these levels. A better understanding of the development of these areas would help to plan SMA 1- tailored supportive programs provided by speech and language therapists, thus enhancing the current recommendations for management in SMA.

DETAILED DESCRIPTION:
Study design: observational longitudinal study. In the first instance, this is intended as a single-centre pilot study with a total duration of 3 years. A larger longitudinal study in a wider national and international cohort will be planned according to preliminary results and insights from this pivotal study. The first appointment will be the screening visit. Initially the trial will be discussed, and informed consent will be obtained for participation in the trial. Information will be collected from the patient and their family including demographics, medical history and detail on medications used by the patient. The investigator will discuss and obtain information on feeding and nutritional support required by the patient, speech and language interventions in place including if they are an augmentative alternative communication user and/or eye tracking device user. After this the investigator will be able to confirm eligibility for the trial. The second visit is the baseline, during this a set of assessments will take place to establish the patients' baseline function. This will include a bulbar function assessment (speech and swallowing), a speech and communication assessment and a cognitive assessment (Thinking abilities; memory, language, reasoning and perception). The investigator will collect further data on respiratory function (breathing) and gross motor function (Muscle strength and abilities). The investigator will assess any adverse events which have occurred since the last visit including symptoms, signs, illness etc. There are further tests which could take place at this visit which are an optional part of the study these include event-related potentials, Brain scan (MRI) and additional communication tests. Patients will then be seen at 6 monthly intervals, at 6m, 12m, 18m, 24m, 30m and 36 months. At each of these appointments and changes to medications will be documented. The investigator will discuss and obtain information on feeding and nutritional support required by the patient, speech and language interventions in place including if they are an augmentative alternative communication user and/or eye tracking device user. Assessments which took place at baseline will be repeated including a bulbar function assessment (speech and swallowing), a speech and communication assessment and we will collect data on respiratory function (breathing) and gross motor function (muscle strength and abilities). Cognitive testing will occur at visits at 12, 24 and 36 months.

At all visits the investigator will assess any adverse events which have occurred since the last visit including symptoms, signs, illness etc. If patients have decided to take part in additional cognitive testing, then this will occur at each 6 monthly visit. The month 36 visit will be the end of study visit so as well as the above will include repeat testing of the optional event-related potentials and brain scan (MRI).

ELIGIBILITY:
Inclusion Criteria:

* genetic documentation of 5q SMA;
* onset of clinical signs and symptoms at ≤ 6 months (180 days) of age;
* 0 - 18 years of age
* treatment with any of the approved disease-modifying therapies;
* parent(s)/legal guardian(s) willing and able to complete the informed consent process and comply with study procedures and visit schedule.

Exclusion criteria:

* any clinically significant medical finding that - in the judgment of the Investigator - will make the patient unsuitable for participation in, and/or unable to complete the study procedures;
* parent(s)/legal guardian(s) unable or unwilling to comply with study procedures and/or refuses to sign consent form.

Exclusion Criteria:

* any clinically significant medical finding that - in the judgment of the Investigator - will make the patient unsuitable for participation in, and/or unable to complete the study procedures;
* parent(s)/legal guardian(s) unable or unwilling to comply with study procedures and/or refuses to sign consent form.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In the first instance, we will recruit SMA 1 paediatric patients (up to 18 years of age) who are under the care of the Neuromuscular team at the Dubowitz Neuromuscular Centre, London, UK, and who are being treated with any approved disease-modifying therapies. A total number of 30 patients is expected to be enrolled in the pilot phase of the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Bulbar function - Changes from baseline | Baseline, Visit Month 12, Month 24, and Months 36
  Paediatric-Functional Oral Intake Scale (p-FOIS/CEDAS)
  Min score( Worse) - Max score 6 (Better performance)
Bulbar function | Visit Month 6
  Paediatric-Functional Oral Intake Scale (p-FOIS/CEDAS)
  Min score 1( Worse) - Max score 6 (Better performance)
Bulbar function | Visit Month 18
  Paediatric-Functional Oral Intake Scale (p-FOIS/CEDAS)
  Min score 1 (Worse) - Max score 6 (Better performance)
Bulbar function | Visit Month 30
  Paediatric-Functional Oral Intake Scale (p-FOIS/CEDAS)
  Min score 1( Worse) - Max score 6 (Better performance)
Speech and Communication - Changes from baseline | Baseline, Month 12, Month 24, and Months 36
  MacArthur-Bates Communicative Development Inventory (MCDI) - Words and Gestures or Words and Sentences
  For 8-18 month-olds looking at words and gestures, the following min score (worse performance) - max scores (better performance) exist:
  Phrases understood: 0/28 Vocabulary understood: 0/396 Vocabulary used: 0/396 Early gestures: 0/18 Later gestures: 0/45 Total gestures: 0/63
  For 18-30 month-olds looking at words and sentences, the following min score (worse performance) - max scores (better performance) exist:
  Words produced = 0/680 Irregular words = 0/25 Overregularized words = 0/45 Sentence complexity = 0/37
Speech and Communication | Visit Month 6
  MacArthur-Bates Communicative Development Inventory (MCDI) - Words and Gestures or Words and Sentences
  For 8-18 month-olds looking at words and gestures, the following min score (worse performance) - max scores (better performance) exist:
  Phrases understood: 0/28 Vocabulary understood: 0/396 Vocabulary used: 0/396 Early gestures: 0/18 Later gestures: 0/45 Total gestures: 0/63
  For 18-30 month-olds looking at words and sentences, the following min score (worse performance) - max scores (better performance) exist:
  Words produced = 0/680 Irregular words = 0/25 Overregularized words = 0/45 Sentence complexity = 0/373
Speech and Communication | Visit Month 18
  MacArthur-Bates Communicative Development Inventory (MCDI) - Words and Gestures or Words and Sentences
  For 8-18 month-olds looking at words and gestures, the following min score (worse performance) - max scores (better performance) exist:
  Phrases understood: 0/28 Vocabulary understood: 0/396 Vocabulary used: 0/396 Early gestures: 0/18 Later gestures: 0/45 Total gestures: 0/63
  For 18-30 month-olds looking at words and sentences, the following min score (worse performance) - max scores (better performance) exist:
  Words produced = 0/680 Irregular words = 0/25 Overregularized words = 0/45 Sentence complexity = 0/37
Speech and Communication | Visit Month 30
  MacArthur-Bates Communicative Development Inventory (MCDI) - Words and Gestures or Words and Sentences
  For 8-18 month-olds looking at words and gestures, the following min score (worse performance) - max scores (better performance) exist:
  Phrases understood: 0/28 Vocabulary understood: 0/396 Vocabulary used: 0/396 Early gestures: 0/18 Later gestures: 0/45 Total gestures: 0/63
  For 18-30 month-olds looking at words and sentences, the following min score (worse performance) - max scores (better performance) exist:
  Words produced = 0/680 Irregular words = 0/25 Overregularized words = 0/45 Sentence complexity = 0/37
Speech and Communication - Changes from baseline | Baseline, Visit Month 6, Month 12, Month 18, Month 24, Month 30 and Months 36
  Peabody Picture Vocabulary Test (PPVT)
Speech and Communication | Visit Month 6
  Peabody Picture Vocabulary Test (PPVT)
  Age-based standard scores (M = 100, SD = 15). Minimum value of normal range is 85, maximum value of normal range is 115, higher score means better outcome.
Speech and Communication | Visit Month 18
  Peabody Picture Vocabulary Test (PPVT)
  Age-based standard scores (M = 100, SD = 15). Minimum value of normal range is 85, maximum value of normal range is 115, higher score means better outcome.
Speech and Communication | Visit Month 30
  Peabody Picture Vocabulary Test (PPVT)
  Age-based standard scores (M = 100, SD = 15). Minimum value of normal range is 85, maximum value of normal range is 115, higher score means better outcome.
Speech and Communication - Changes from Baseline | Baseline, Month 12, Month 24, and Months 36
  Social Communication Questionnaire (SCQ)
  Minimum value is 0, maximum value is 39, higher score means worse outcome (The threshold varies depending on countries and researchers).
Speech and Communication | Visit Month 6
  Social Communication Questionnaire (SCQ)
  Minimum value is 0, maximum value is 39, higher score means worse outcome (The threshold varies depending on countries and researchers).
Speech and Communication | Visit Month 18
  Social Communication Questionnaire (SCQ)
  Minimum value is 0, maximum value is 39, higher score means worse outcome (The threshold varies depending on countries and researchers).
Speech and Communication | Visit Month 30
  Social Communication Questionnaire (SCQ)
  Minimum value is 0, maximum value is 39, higher score means worse outcome (The threshold varies depending on countries and researchers).

SECONDARY OUTCOMES:
Cognitive function - Changes from baseline | Baseline, Month 12, Month 24, and Months 36
  Bayley Scales of Infant & Toddler Development - Forth Edition
  Age-based standard scores (M = 100, SD = 15). Minimum value of normal range is 85, maximum value of normal range is 115, higher score means better outcome.
Cognitive function | Visit Month 6
  Bayley Scales of Infant & Toddler Development - Forth Edition
  Age-based standard scores (M = 100, SD = 15). Minimum value of normal range is 85, maximum value of normal range is 115, higher score means better outcome.
Cognitive function | Visit Month 18
  Bayley Scales of Infant & Toddler Development - Forth Edition
  Age-based standard scores (M = 100, SD = 15). Minimum value of normal range is 85, maximum value of normal range is 115, higher score means better outcome.
Cognitive function | Visit Month 30
  Bayley Scales of Infant & Toddler Development - Forth Edition
  Age-based standard scores (M = 100, SD = 15). Minimum value of normal range is 85, maximum value of normal range is 115, higher score means better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No